CLINICAL TRIAL: NCT05368831
Title: A Phase 1, Open-label Study to Evaluate the Effects of NST-1024 on the Pharmacokinetics of Caffeine, Flurbiprofen, Omeprazole, Metoprolol, and Midazolam in Healthy Subjects
Brief Title: Open-label Study to Evaluate the Effects of NST-1024 on the PK of Multiple Drugs in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NST-1024-02
Record Dates: First submitted 2022-04-29; First posted 2022-05-10 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral dose of NST-1024, Caffeine, Flurbiprofen, Omeprazole, Metoprolol, and Midazolam (Experimental): Day 1: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam
  * Days 8 to 22: oral doses of 200 mg NST-1024 qd multiple-dose regimen
  * Day 8: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024
  * Day 21: single oral dose of 100 mg caffeine and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024.
  Interventions: Drug: NST-1024

INTERVENTIONS:
Drug: NST-1024 — Drug Drug interactions between NST-1024 and caffeine (and paraxanthine), flurbiprofen, omeprazole, metoprolol, and midazolam

SUMMARY:
Phase 1, open label study to evaluate the effects of NST-1024 on the pharmacokinetics (PK) of caffeine (and paraxanthine), flurbiprofen, omeprazole, metoprolol, and midazolam (and 1-hydroxymidazolam) in healthy male and female subjects.

DETAILED DESCRIPTION:
Up to 21 subjects will be enroled to ensure that 18 subjects complete the study. All subjects will receive each of the following treatments:

* Day 1: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam
* Days 8 to 22: oral doses of 200 mg NST-1024 qd multiple-dose regimen
* Day 8: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024
* Day 21: single oral dose of 100 mg caffeine and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 65 years of age, inclusive.
2. Body mass index between 18.0 and 32.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhaemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and/or check in and from the physical examination at check-in, as assessed by the investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in Appendix 4.
5. Able to comprehend and willing to sign an Informed Consent Form (ICF) and to abide by the study restrictions

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular (CV), gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of febrile illness within 1 week prior to the first dose.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
* Confirmed (eg, 2 consecutive measurements) systolic blood pressure >160 or <80 mmHg, diastolic blood pressure >90 or <45 mmHg, and pulse rate >100 or <40 beats per minute.
* Positive hepatitis panel and/or positive human immunodeficiency virus test
* Administration of a coronavirus disease 2019 vaccine in the past 30 days prior to dosing.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including over-the-counter and herbal medication, within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the investigator (or designee).
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
* Alcohol consumption of >21 units (males) and >14 units (females) per week. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
* Receipt of blood products within 2 months prior to check in.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following screening, eligible participants were to receive each of the following treatments:
  * Day 1: Probe Drugs Cocktail #1
  * Day 8: 200 mg NST-1024 + Probe Drug Cocktail #1
  * Days 8 to 22: 200 mg NST-1024 once daily
  * Day 21: 200 mg NST-1024 + Probe Drug Cocktail #2
Groups:
- All Treated Participants: All participants received each of the following treatments:
  * Day 1: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam
  * Day 8: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024
  * Days 8 to 22: oral doses of 200 mg NST-1024 qd multiple-dose regimen
  * Day 21: single oral dose of 100 mg caffeine and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024.
Period: Probe Drugs Cocktail #1
Arm/Group | All Treated Participants
Started | 24
Completed | 24
Not Completed | 0
Period: 200 mg NST-1024 + Probe Drug Cocktail #1
Arm/Group | All Treated Participants
Started | 24
Completed | 24
Not Completed | 0
Period: 200 mg NST-1024 (QD)
Arm/Group | All Treated Participants
Started | 24
Completed | 21
Not Completed | 3
Not completed — Adverse Event | 3
Period: 200 mg NST-1024 (QD) + Probe Cocktail #2
Arm/Group | All Treated Participants
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated Participants: * Day 1: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam
  * Days 8 to 22: oral doses of 200 mg NST-1024 qd multiple-dose regimen
  * Day 8: single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024
  * Day 21: single oral dose of 100 mg caffeine and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Effects of NST-1024 on the AUC0-t vs Time of Caffeine, Flurbiprofen, Omeprazole, Metoprolol, and Midazolam in Healthy Male and Female Subjects
Description: Evaluate the effects of NST-1024 on the pharmacokinetics (PK) (AUC0-t) of caffeine, flurbiprofen, omeprazole, metoprolol, and midazolam in healthy male and female subjects
Time Frame: 15 days
Population: PK analysis population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Probe Drugs Cocktail #1: Participants received a single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam on day 1. Each dose was administered with approximately 240 mL of room temperature water, though additional water (up to another approximately 240 mL) was permissible. All doses were given in a fasted state.
- 200 mg NST-1024 + Probe Drug Cocktail #1: Participants received a single oral dose of 100 mg caffeine, 50 mg flurbiprofen, 20 mg omeprazole, 100 mg metoprolol, and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024 on day 8. Each dose was administered with approximately 240 mL of room temperature water, though additional water (up to another approximately 240 mL) was permissible. All doses were given in a fasted state.
- 200 mg NST-1024 (QD) + Probe Drugs Cocktail #2: Participants received a single oral dose of 100 mg caffeine and 2.5 mg midazolam coadministered with an oral dose of 200 mg NST-1024 on day 21. Each dose was administered with approximately 240 mL of room temperature water. All doses were given in a fasted state.
Arm/Group | Probe Drugs Cocktail #1 | 200 mg NST-1024 + Probe Drug Cocktail #1 | 200 mg NST-1024 (QD) + Probe Drugs Cocktail #2
Number analyzed (Participants) | 23 | 23 | 21
h*ng/mL
  Caffeine: number analyzed (Participants) | 19 | 19 | 21
  Caffeine | 17100 (44.5) | 17100 (43.4) | 17200 (39.1)
  Paraxanthine: number analyzed (Participants) | 16 | 12 | 21
  Paraxanthine | 10300 (29.4) | 9920 (33.9) | 10500 (35.6)
  Midazolam: number analyzed (Participants) | 21 | 21 | 21
  Midazolam | 35.3 (39.5) | 37.9 (28.2) | 33.0 (43.4)
  1-Hydroxymidazolam: number analyzed (Participants) | 21 | 21 | 21
  1-Hydroxymidazolam | 9.99 (44.7) | 10.3 (50.4) | 11.6 (24.7)
  Flurbiprofen: number analyzed (Participants) | 21 | 21 | 0
  Flurbiprofen | 37600 (27.3) | 34500 (29.4) |
  Metoprolol: number analyzed (Participants) | 21 | 21 | 0
  Metoprolol | 654 (89.0) | 745 (75.0) |
  Omeprazole: number analyzed (Participants) | 20 | 20 | 0
  Omeprazole | 428 (120.8) | 432 (140.9) |

2. Primary Outcome: Evaluate the Effects of NST-1024 on the Plasma Concentration (Cmax) of Caffeine, Flurbiprofen, Omeprazole, Metoprolol, and Midazolam in Healthy Male and Female Subjects
Description: Evaluate the effects of NST-1024 on the PK (Cmax) of caffeine, flurbiprofen, omeprazole, metoprolol, and midazolam in healthy male and female subjects
Time Frame: 15 days
Population: PK analysis population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Probe Drugs Cocktail #1 | 200 mg NST-1024 + Probe Drug Cocktail #1 | 200 mg NST-1024 (QD) + Probe Drugs Cocktail #2
Number analyzed (Participants) | 23 | 23 | 21
ng/mL
  Caffeine: number analyzed (Participants) | 19 | 19 | 21
  Caffeine | 2390 (21.9) | 2390 (26.4) | 2330 (25.4)
  Paraxanthine: number analyzed (Participants) | 16 | 12 | 21
  Paraxanthine | 656 (18.8) | 630 (17.5) | 617 (20.4)
  Midazolam: number analyzed (Participants) | 21 | 21 | 21
  Midazolam | 12.8 (26.8) | 12.8 (24.7) | 12.1 (35.0)
  1-Hydroxymidazolam: number analyzed (Participants) | 21 | 21 | 21
  1-Hydroxymidazolam | 4.14 (46.7) | 3.69 (63.5) | 4.54 (37.1)
  Flurbiprofen: number analyzed (Participants) | 21 | 21 | 0
  Flurbiprofen | 7240 (32.9) | 6480 (36.4) |
  Metoprolol: number analyzed (Participants) | 21 | 21 | 0
  Metoprolol | 127 (53.0) | 142 (58.6) |
  Omeprazole: number analyzed (Participants) | 21 | 21 | 0
  Omeprazole | 221 (86.9) | 189 (115.5) |

3. Secondary Outcome: Assess Adverse Event (AEs) and Serious Adverse Event (SAEs) to Determine Safety Profile of NST-1024 in Healthy Subjects
Description: Assess AEs and SAEs to support ongoing safety profile data
Time Frame: 15 days
Measure: Number; unit: participants
Groups:
- 200 mg NST-1024 (QD): Participants received oral doses of 200 mg NST-1024 on study days 8-22. Each dose was administered with approximately 240 mL of room temperature water
Arm/Group | Probe Drugs Cocktail #1 | 200 mg NST-1024 + Probe Drug Cocktail #1 | 200 mg NST-1024 (QD) | 200 mg NST-1024 (QD) + Probe Drugs Cocktail #2
Number analyzed (Participants) | 24 | 24 | 24 | 21
participants
  Overall | 6 | 6 | 9 | 8
  Serious | 0 | 0 | 0 | 0
  Leading to discontinuation | 0 | 0 | 3 | 0
  Leading to death | 0 | 0 | 0 | 0
  Severity - Mild | 6 | 6 | 9 | 7
  Severity - Moderate | 0 | 0 | 0 | 2
  Severity - Severe | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening to up to 10 days post final dose follow up, approximately 2 months.
Description: Whilst only 24 participants were enrolled in total, the different treatment regimens administered have been displayed as different arms/ groups to allow comparison of results between the different treatments.
Arm/Group | Probe Drugs Cocktail #1 | 200 mg NST-1024 + Probe Drug Cocktail #1 | 200 mg NST-1024 (QD) | 200 mg NST-1024 (QD) + Probe Drugs Cocktail #2
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 6/24 | 6/24 | 9/24 | 8/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Probe Drugs Cocktail #1 (N=24) | 200 mg NST-1024 + Probe Drug Cocktail #1 (N=24) | 200 mg NST-1024 (QD) (N=24) | 200 mg NST-1024 (QD) + Probe Drugs Cocktail #2 (N=21)
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Application site erythema (General disorders) | 1 | 1 | 0 | 0
Catheter site swelling (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT05368831/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05368831/SAP_001.pdf